CLINICAL TRIAL: NCT03559868
Title: Inhibition of Sterile Inflammation by Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2000025289; 1U01AA026962-01 (NIH)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Response
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Digoxin 3 mcg/Kg/day (Active Comparator): Patients receiving oral digoxin 3 mcg/Kg/day
  Interventions: Drug: Digoxin
- Digoxin 0.15 mcg (Active Comparator): Patients receiving oral digoxin 0.15 mcg/Kg/day
  Interventions: Drug: Digoxin
- Placebo (Placebo Comparator): oral placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Digoxin — Participants will receive 3 mcg/Kg/day doses of oral digoxin
  Arms: Digoxin 3 mcg/Kg/day
Other: Placebo — Oral placebo
  Arms: Placebo
Drug: Digoxin — Participants will receive 0.15 mcg/Kg/day doses of oral digoxin
  Arms: Digoxin 0.15 mcg

SUMMARY:
To investigate the effect of digoxin on pyruvate kinase isoform 2 (PKM2) binding to pro-inflammatory loci and innate immune inflammatory responses in the peripheral blood in healthy subjects.

DETAILED DESCRIPTION:
To investigate the effect of orally administered digoxin on innate immune inflammatory responses in the peripheral blood of healthy subjects. We hypothesize the reduction in innate immune inflammatory responses will be expected in the peripheral blood with the effect of oral digoxin.

To investigation how human peripheral blood immune cells change their inflammatory responses after exposure to digoxin in vitro.

ELIGIBILITY:
Inclusion Criteria

1. Age >18 y ≤ 70 years
2. subjects with normal serum creatinine, normal EKG and currently not taking any medication.

Exclusion criteria

1. Autoimmune liver disease (ANA > 1/320)
2. Chronic viral hepatitis
3. Hepatocellular carcinoma
4. Complete portal vein thrombosis
5. Extrahepatic terminal disease
6. Pregnancy
7. Treatment with prednisolone or pentoxifyllin for more than 3 days prior to inclusion/start date
8. Active alcohol abuse (>50 g/day for men and >40 g/day for women) in the last 3 months
9. AST > ALT and total bilirubin > 3 mg/dl in the past 3 months
10. Liver biopsy and/or clinical picture consistent with alcoholic hepatitis
11. Lack of signed informed consent.
12. Known hypersensitivity to digoxin or other forms of digitalis, ventricular fibrillation.
13. Any significant medical conditions, any electrolyte abnormalities, over the counter medications, natural products and prescription drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wajahat Mehal, MD, Principal Investigator — Yale University
Locations (1):
- Yale Centre of Clinical Investigation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were consented but never started.
Period: Overall Study
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
Started | 14 | 14 | 14
Completed | 6 | 6 | 7
Not Completed | 8 | 8 | 7

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only collected from completers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9) | 31.3 (15) | 37.7 (12) | 36.1 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 14
  Male | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 3
  White | 4 | 6 | 1 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Lower Levels of Spontaneous Reactive Oxygen Species (ROS) Production
Description: Investigators will be take neutrophils (PMN's) from the blood and seeing if the patients on digoxin have lower levels of spontaneous reactive oxygen species (ROS) production. This will be determined as a greater than 25% reduction in ROS compared to individuals not taking digoxin. The serum digoxin levels are just being done per usual guidelines to make sure that supratherapeutic levels of digoxin are not reached.
Time Frame: after starting digoxin
Population: No data for this outcome was collected.
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Lower Levels of Spontaneous Reactive Oxygen Species (ROS) Production
Description: Investigators will take neutrophils (PMN's) from the blood and seeing if the patients on digoxin have lower levels of spontaneous reactive oxygen species (ROS) production. This will be determined as a greater than 25% reduction in ROS compared to individuals not taking digoxin. The serum digoxin levels are just being done per usual guidelines to make sure that supratherapeutic levels of digoxin are not reached.
Time Frame: 1 week after starting digoxin
Population: No data for this outcome was collected.
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Lower Levels of Spontaneous Reactive Oxygen Species (ROS) Production
Description: as for outcome 2
Time Frame: 2 weeks after starting digoxin
Population: No data for this outcome was collected.
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Lower Levels of Spontaneous Reactive Oxygen Species (ROS) Production
Description: as for outcome 2
Time Frame: 3 weeks after starting digoxin
Population: No data for this outcome was collected.
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Investigation of How Human Peripheral Blood Immune Cells Change Their Inflammatory Responses After Exposure to Digoxin in Vitro
Description: Blood (25ml) will be obtained from healthy blood donors at one time. Human peripheral monocytes will be isolated using Polymorphprep™ density sedimentation according to the manufacturer's instructions. Data presented here are the mean concentrations.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
Number analyzed (Participants) | 6 | 6 | 7
pg/ml
  CCL2 | 697 (237) | 1351 (483) | 5790 (2442)
  CCL4 | 1205 (569) | 12180 (9763) | 22328 (7251)
  CCL20 | 894 (490) | 1205 (569) | 1761 (471)
  CXCL1 | 312 (232) | 1437 (340) | 2909 (725)
  CXCL10 | 366 (293) | 2472 (886) | 4452 (1549)
  G-CSF | 35 (19) | 211 (80) | 323 (129)
  GM-CSF | 42 (15) | 142 (39) | 231 (60)
  Granzyme B | 182 (60) | 1117 (684) | 2734 (1582)
  IFN Alpha | 26 (31) | 97 (61) | 174 (109)
  IFN Gamma | 27 (9) | 103 (82) | 229 (99)
  IL-RA | 1074 (290) | 6040 (1785) | 12618 (3485)
  IL-6 | 1064 (427) | 2797 (831) | 5006 (1171)
  PDGF AA | 238 (294) | 1519 (773) | 2848 (135)
  PDGF AB/BB | 128 (75) | 908 (539) | 1038 (587)
  TNF Alpha | 173 (92) | 2786 (956) | 4040 (1004)
  IL-8 | 117 (41) | 306 (52) | 420 (24)
  Galactin 9 | 11977 (4287) | 20623 (5876) | 25999 (2645)
  IL10 | 26069 (6793) | 17528 (9660) | 2300 (2230)
Statistical Analysis 1: Comparison: Digoxin 3 mcg/Kg/Day vs Digoxin 0.15 mcg; For IL10; Test type: Superiority; p < 0.01, ANOVA; Ordinary one-way ANOVA Bartlett's test

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Digoxin 3 mcg/Kg/Day | Digoxin 0.15 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03559868/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT03559868/ICF_000.pdf